CLINICAL TRIAL: NCT00299286
Title: A Double Blind Short-Term Presurgical Study Assessing the Molecular Antiproliferative Predictors of Lapatinib's Effects in Breast Cancer
Brief Title: Short-term Presurgical Study to Assess Molecular Predictors of Lapatinib's Effects in Primary Breast Cancer
Acronym: MAPLE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCR2737
Record Dates: First submitted 2006-03-03; First posted 2006-03-06 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-08

CONDITIONS: Breast Cancer
Keywords: Ki67; Molecular; antiproliferative
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lapatinib (Experimental): lapatinib oral 1500mg daily taken as 6 tablets as one dose 10-14 days presurgery
  Interventions: Drug: Lapatinib
- Lapatinib-Placebo (Placebo Comparator): placebo comparator 6 tablets taken as one dose daily
  Interventions: Drug: Lapatinib-Placebo

INTERVENTIONS:
Drug: Lapatinib — In order for patients to take their study medication for 14 days only, treatment should commence on the 14th day prior to the day before scheduled surgery (i.e. if surgery is scheduled for the 15th of the month, tablets should be taken from the 1st to the 14th of that month).
  Lapatinib tablets are dispensed as 250mg tablets. Patients should be advised to take all 6 tablets at once as one dose (total daily dose 1500mg). Tablets should be taken on an empty stomach either one hour before or one hour after a meal at the same time each day and according to the instructions on the bottle.
  Other Names: Tyverb
  Arms: Lapatinib
Drug: Lapatinib-Placebo — In order for patients to take their study medication for 14 days only, treatment should commence on the 14th day prior to the day before scheduled surgery (i.e. if surgery is scheduled for the 15th of the month, tablets should be taken from the 1st to the 14th of that month).
  Lapatinib-placebo tablets will be composed of lactose, cellulose, starch, magnesium stearate, and coated with Opadryl orange and look the same as the active treatment. The patients should take all 6 tablets at once as one dose.
  Arms: Lapatinib-Placebo

SUMMARY:
To provide an in vivo measure of the activity of lapatinib. To assess the antiproliferative effects of lapatinib in breast cancer, ie how much lapatinib slows down the growth of cancer cells by measuring K167 (a marker of proliferation) in breast tumours before and after a short treatment with lapatinib.

DETAILED DESCRIPTION:
Randomised multi centre double blind pre-surgical study in women with a histological diagnosis of breast cancer by core biopsy.

ELIGIBILITY:
Inclusion Criteria:

Patients must have a histological or cytologic diagnosis of primary breast cancer with a tumour size adequate for multiple core biopsies Informed signed consent Scheduled for primary surgery Expected to be compliant for duration of study Age<80 ECOG performance status 0-2 (Karnofsky >60%) Cardiac ejection fraction within the institutional range of normal as measured by echocardiogram or MUGA scan Eligibility of patients receiving medications known to affect, or with the potential to affect the activity or pharmacokinetics of lapatinib will be determined following review by the Trial Coordinator The effects if lapatinib on the developing fetus are unknown. For this reason, women of childbearing potential must agree to use adequate non-hormonal contraception for the duration of study participation.

Able to swallow and retain oral medication.

Exclusion Criteria:

Patients with prior diagnosis of malignancy except in situ disease or basal cell carcinoma of the skin.

Patients may be receiving any other investigational agents or receiving concurrent anticancer therapy. In addition, all herbal (alternative) medicines are excluded.

Evidence of metastatic disease. Use of hormonal therapy such as oral contraceptives or hormonal replacement therapy within 4 weeks of study entry.

Regular use of steroid hormones or other agents that could influence study endpoints History of allergic reactions attributed to compounds of similar chemical or biologic composition to GW572016.

Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/ social situations that would limit compliance with study requirements.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2007-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Changes in Ki67 after short term treatment with lapatinib. | 11-14 days after treatment
  Paired core samples taken at baseline and time of main surgery analysed for Ki67, TUNEL, HER2, EGFR, ER, PgR, pAkt,pERK & stathmin

SECONDARY OUTCOMES:
Assess how changes in Ki67 and apoptosis relate to molecular markers at baseline and after 2 weeks. These markers aer HER2, EGFR, p-HER2, p-EGFR, p-ERK1/2, pAKT, ER, PR, IGR-1R, cyclin D1, PTEN and TGF alpha. Further markers may be considered. | 10-14 days after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Professor Ian Smith, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden NHS Foundation Trust, London, United Kingdom